CLINICAL TRIAL: NCT04523168
Title: A Phase II Study Testing the Feasibility and Efficacy of Coronary Sinus Narrowing in Patients With Coronary Microvascular Dysfunction
Brief Title: Feasibility and Efficacy of Coronary Sinus Narrowing in Patients With Coronary Microvascular Dysfunction
Acronym: Reducer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amir Lerman (Other)
Responsible Party: Sponsor-Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-006386
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Coronary Microvascular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Chronic Refractory Angina (Experimental): Subjects with chronic refractory angina will undergo implantation of the Neovasc Reducer™ System in the cardiac catheterization laboratory.
  Interventions: Device: The Neovasc Reducer™ System

INTERVENTIONS:
Device: The Neovasc Reducer™ System — A stainless-steel mesh pre-mounted on a customized hourglass shaped balloon catheter, is designed to create a focal narrowing in the lumen of the CS to generate a pressure gradient across it.

SUMMARY:
This study is being done to evaluate the role of a novel implantable device, called The Neovasc Reducer™ System, in improving microvascular function, symptoms and quality of life in symptomatic patients with coronary microvascular dysfunction.

ELIGIBILITY:
Inclusion Criteria

* Age >18
* Able to provide written informed consent and willing to participate in all required study follow-up assessments
* Symptomatic CAD with refractory angina defined as CCS class II to IV, despite optimal tolerated medical therapy
* Abnormal coronary microvascular function indices: CFR≤2.5 and/or IMR≥25

Exclusion Criteria

* Recent (within 3 months) acute coronary syndrome
* Patients with prior coronary artery bypass surgery
* Unstable angina (recent onset angina, crescendo angina, or rest angina with ECG changes) during the last 30 days
* Subjects in cardiogenic shock (systolic pressure < 80mm/Hg, on vasopressors or intraaortic counter pulsation) at the time of consenting. Subjects who recover from cardiogenic shock by the time of consenting are eligible.
* Obstructive CAD on coronary angiography (>70% stenosis or 50-70% stenosis with iFR<0.89 or FFR<0.8 in epicardial artery)
* Inability to perform invasive coronary flow evaluation and/or measure CFR and IMR in the LAD
* Severe valvular heart disease
* LVEF<30%
* Decompensated congestive heart failure (CHF) or hospitalization due to CHF during the last 3 months
* Patient with a pacemaker electrode in the CS
* Mean right atrial pressure >15 mmHg
* Anomalous or abnormal CS anatomy (e.g., tortuosity, aberrant branch, persistent left superior vena cava (SVC) as demonstrated on angiogram
* CS diameter at the site of planned implantation greater than 13mm or less than 9.5 mm as measured by angiogram
* Severe chronic obstructive pulmonary disease (COPD) indicated by a forced expiratory volume in one second that is less than 55 percent of the predicted value
* Tricuspid valve replacement or repair (tissue or mechanical)
* Chronic renal failure (serum creatinine >2mg/dL), and or on chronic hemodialysis
* Moribund, or with comorbidities limiting life expectancy to less than one year
* Known severe reaction to required procedural medication
* Known allergy to stainless steel or nickel
* Magnetic Resonance Imaging (MRI) within 8 weeks of Reducer implantation
* Participation in another ongoing investigational trial
* Additional factors deemed unsuitable for trial enrollment per discretion of principal investigator
* Inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Refractory Angina
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Refractory Angina
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Coronary Flow Reserve (CFR)
Description: Coronary flow reserve is calculated as the ratio of hyperemic or maximal flow down a coronary vessel to the resting coronary blood flow.
Time Frame: Baseline, 120 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Chronic Refractory Angina
Number analyzed (Participants) | 30
ratio | 3.04 (1.06)
Statistical Analysis 1: Comparison: Chronic Refractory Angina; Baseline, 120 days; Test type: Superiority; p = 0.0137, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Seattle Angina Questionnaire (SAQ)
Description: The Seattle Angina Questionnaire (SAQ) is a self-administered, 19-item questionnaire with 5 different subscales - physical limitations, angina stability, angina frequency, treatment satisfaction and quality of life. Each subscale score ranges from 0 to 100, where higher scores indicate better health outcomes.
Time Frame: 120 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Refractory Angina
Number analyzed (Participants) | 30
score on a scale
  Physical limitation score | 62.4 (26.8)
  Angina stability score | 67.5 (28.7)
  Angina frequency score | 49.9 (31.3)
  Treatment satisfaction score | 81.2 (17.3)
  Quality of life score | 54.7 (28.4)

3. Secondary Outcome: Change in Canadian Cardiovascular Society (CCS) Angina Class
Description: The Canadian Cardiovascular Society (CCS) Angina Class symptom scale classifies anginal symptoms. Scores range from 1 (best; everyday, regular, physical activity does not cause angina) to 4 (worst; unable to do any regular physical activity without discomfort, anginal symptoms may be present at rest).
Time Frame: Baseline, 120 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Refractory Angina
Number analyzed (Participants) | 30
score on a scale | 2.40 (1.10)
Statistical Analysis 1: Comparison: Chronic Refractory Angina; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from time of enrollment through four months following device implant, for a total of approximately five months.
Arm/Group | Chronic Refractory Angina
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Refractory Angina (N=30)
Wire related perforations (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Refractory Angina (N=30)
Vomiting/Nausea/Reflux (Gastrointestinal disorders) | 7 (10)
Headache (General disorders) | 4 (4)
Shortness of breath (General disorders) | 3 (7)
Fever/chills/diarrhea (General disorders) | 1 (1)
Infection (Infections and infestations) | 6 (6)
General joint pain (General disorders) | 8 (9)
Lightheaded/dizzy/sycope (General disorders) | 4 (4)
Chest pain (Cardiac disorders) | 7 (9)
Bruising (General disorders) | 3 (3)
Inflammation (General disorders) | 3 (3)
Irregular heart rate (Cardiac disorders) | 4 (4)
Low blood pressure (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT04523168/Prot_SAP_000.pdf